CLINICAL TRIAL: NCT05253014
Title: Comparative Study Between Different Approaches for the Management of Post-dural Puncture Headache
Brief Title: Different Approaches for the Management of Post-dural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahaa Mohammed Refaie (Other)
Responsible Party: Sponsor-Investigator, Bahaa Mohammed Refaie, lecturer of anesthesia and ICu, Sohag University
Organization: Sohag University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2223
Record Dates: First submitted 2022-02-05; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lidocaine group (Active Comparator)
  Interventions: Procedure: sphenopalatine ganglion block
- bupivacaine group (Active Comparator)
  Interventions: Procedure: sphenopalatine ganglion block
- conservative group (Active Comparator)
  Interventions: Drug: paracetamol

INTERVENTIONS:
Procedure: sphenopalatine ganglion block — block of the sphenopalatine ganglion using either lidocaine or bupivacaine to relief postdural puncture headache
  Arms: bupivacaine group; lidocaine group
Drug: paracetamol — intravenous paracetamol every 8 hours
  Arms: conservative group

SUMMARY:
Detecting the efficacy and safety of trans-nasal sphenopalatine ganglion block using either lidocaine 2% or bupivacaine 0.5 % as a treatment line for post-dural puncture headache

ELIGIBILITY:
Inclusion Criteria:

* The ASA physical condition І-П
* the patient underwent CS under spinal anesthesia
* The headache developed within 5 days after the dural puncture
* There is no different explanation for the headache

Exclusion Criteria:

* coagulopathy
* history of nasal bleeding
* nasal polyp
* septal deviation
* local anesthetics reaction

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 20 - 45 years old female with PDPH after cesarean section using spinal anesthesia
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
postdural puncture headache | within five days after the dural puncture
  visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided